CLINICAL TRIAL: NCT03192501
Title: Multicentre Perspective Non-interventional Study of Survival Benefits of iCAGES-guided Therapy in Contrast to Standard Therapy or IHC-guided Therapy for Advanced Cancers
Brief Title: iCAGES-guided Precision Therapy for Cancers in Contrast to Standard Care or IHC-guided Theray
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZZiCAGES-001
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Gene Abnormality; Gene Product Sequence Variation; Cancer
Keywords: lung cancer; iCAGES; gene mutation; precision medicine; advanced cancers; IHC; Targeted therapy
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Erlotinib Hydrochloride; capmatinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — cancer biopsy samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Study group (A group): In this group, we perform whole exome or genome sequencing of tumor sample in compared to blood sample, screen tumor-related special mutations by using biomedical informatics analysis procedure and utilized the iCAGES system to rank the most appropriate drugs available and then manually examine this list to select the best therapeutic strategy for the patient based on availability of drug and expert knowledge. The PFS, OS, and quality of life (QOL) will be recorded and compared with that from standard care.
  Interventions: Drug: inhibitors, ADC drugs such as tarceva, capmatinib, padcev et al for A/C group.
- Control group (B group): In this group, patients with advanced cancers (matched with Group A) will be treated under the guidance of NCCN, without performing iCAGES analysis.
- Control group (C group): In this group, patients with advanced cancers (matched with Group A) will be treated with appropriate targeted drugs according to IHC detection of more than 20 protein molecules with blank tissue slides from the cancer.
  Interventions: Drug: inhibitors, ADC drugs such as tarceva, capmatinib, padcev et al for A/C group.

INTERVENTIONS:
Drug: inhibitors, ADC drugs such as tarceva, capmatinib, padcev et al for A/C group. — Choose appropriate targeted drugs according to NGS/IHC results.
  Groups: Control group (C group); Study group (A group)

SUMMARY:
This study prospectively evaluates whether the use of iCAGES (integrated CAncer GEnome Score) tool in guiding the treatment of advanced cancers is superior to current standard care or IHC-guided therapy in progress free survival (PFS),overall survival (OS),and improvement of life quality.

DETAILED DESCRIPTION:
Cancer is a fatal disease caused by the accumulation of various oncogene and tumor suppressor gene mutations. Studies of high-throughput sequencing for patients who suffered from cancer has found that different mutations play a different role in the occurrence and development of different cancers. Several gene panels already exist to help identify mutations in a few genes that may have corresponding FDA-approved drugs or drugs under clinical trials. However, given whole-genome/exome sequencing data, the suitable clinical analysis tool to analyze individualized cancer-related gene mutations, and recommend the most appropriate targeted treatment options among hundreds of possible drugs therapy is absent currently.

The recently proposed iCAGES is a precise biomedical informatics analysis tool, which could help increase the accuracy of cancer driver gene detection and prioritization, bridge the gap between personal cancer genomic data and prior cancer research knowledge,and facilitate cancer molecular diagnosis as well as personalized precision therapy.

IHC detection of multiple molecules such as EGFR, HER2-3, TROP3, NECTIN4, MET, B7-H3-4, B1-H7, Claudin18.2, FGFR1-4, Mesothelin, ROR1, BCMA, AXL, TF, FRα, CD70, PPARα, HIF-2α, RET, ROS1, NTRK, CDK4/6, FLT3, EZH2 are also scheduled for appropriate targeted therapy and comparison if available.

ELIGIBILITY:
Inclusion Criteria:

* Pathological and clinical diagnosis of recurrence / metastatic lung cancer or other advanced cancers.
* There are PACS images available at the Second Affiliated Hospital of Guangzhou Medical University and the collaborated Hospitals.
* The patient is informed consent and signed a written consent.

Exclusion Criteria:

* Age > 70 or <18 years old.
* Previous history of malignant tumors.
* Pregnant or lactating female patients.
* Any serious concomitant disease that is expected to have an adverse effect on prognosis, including the heart disease that treatment is required, unsatisfactory controlled diabetes and psychiatric disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, all the patients will be recruited from the Second Affiliated Hospital of Guangzhou Medical University and the collaborated Hospitals during 01/07/2017 to 01/07/2019, 250 advanced patients (90 cases for A group, 70 cases for B group, and 90 cases for C group) are anticipated to be collected. All the patients are more than 18 years old and less than 75 years old. The follow-up will be performed every 2 month until 2 years after the first treatment post-recruitment or quit.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2039-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  The PFS will be recorded during the follow up time.
OS | 2 years
  The OS will be recorded during the follow up time.

SECONDARY OUTCOMES:
Quality of life. | 2 years
  Physicians Global Assessment to measure quality of life
Pain | one year
  Visual Analog Score for pain

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong C, Guo Y, Yang H, He Z, Liu X, Wang K. iCAGES: integrated CAncer GEnome Score for comprehensively prioritizing driver genes in personal cancer genomes. Genome Med. 2016 Dec 22;8(1):135. doi: 10.1186/s13073-016-0390-0. PMID 28007024
- See also: test link — http://nih.gov